CLINICAL TRIAL: NCT00041509
Title: ThromboEMbolism Prevention Efficacy and Safety Trial (TEMPEST): A Double-blind Four-week Study to Assess the Efficacy, Safety, and Tolerability of SB-424323 in the Extended Prophylaxis of Patients Following Total Hip Arthroplasty
Brief Title: ThromboEmbolism Prevention Efficacy and Safety Trial (TEMPEST)
Acronym: TEMPEST
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 424323/025
Record Dates: First submitted 2002-07-09; First posted 2002-07-12 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Arthroplasty
Keywords: venous thromboembolism; thromboembolism; pulmonary embolism; deep vein thrombosis
MeSH Terms: conditions — Venous Thromboembolism; Thromboembolism; Pulmonary Embolism; Venous Thrombosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- SB424323, 500 mg BID (Experimental)
  Interventions: Drug: SB-424323
- SB424323, 125 mg BID (Experimental)
  Interventions: Drug: SB-424323
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SB-424323 — 500 mg, oral, BID for 28 days or 125 mg, oral, BID for 28 days
  Arms: SB424323, 125 mg BID; SB424323, 500 mg BID
Drug: Placebo — matching placebo, oral, BID for 28 days
  Arms: Placebo

SUMMARY:
The purpose of this study is to gain additional safety information as well as to determine after the study drug has been given to patients who have undergone total hip replacement surgery, whether the study drug is effective in preventing late deep vein thrombosis (blood clots in legs) or pulmonary embolism (blood clots in lungs).

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for primary elective unilateral total hip arthroplasty (i.e. first time the hip is being replaced on the operative side).
* Patients who have given written informed consent to participate in this study.

Exclusion Criteria:

* Patients with a contraindication to contrast venography
* Patients with an increased risk of bleeding.
* Patients with a predefined risk for prethrombotic episodes or a history of thrombophilia.
* Other inclusion or exclusion criteria to be determined by the physician and study sponsor.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 343 (Actual)
Dates: Start 2002-01; Primary Completion 2003-05 (Actual); Study Completion 2003-05 (Actual)

PRIMARY OUTCOMES:
VTE | 28 day treatment period
  Incidence of VTE during the 28-day treatment period, including death due to VTE

SECONDARY OUTCOMES:
types of VTE | 28 day treatment period
  The incidence of the types of VTE including, DVT (deep vein thrombosis), symptomatic VTE, PE] and anti-IIa activity

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline